CLINICAL TRIAL: NCT06928441
Title: Non-invasive Vagus Nerve Stimulation and Sleep in Healthy Volunteers: a Randomized Trial.
Brief Title: Non-invasive Vagus Nerve Stimulation and Sleep in Healthy Volunteers.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: REB24-1438
Record Dates: First submitted 2025-04-01; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Sleep
Keywords: Neuromodulation, Vagus nerve

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trial Arm 1 (Experimental): Participants and experimenters are blinded. The aim of this study is to determine whether a battery-operated portable device (current adjustable) attached to the outer ears (tragus) makes one more likely to improve on their sleep and quality of daily life. Investigators believe this device encourages increases in vagal tone associated with increases in baroreflex sensitivity, improving sleep and possibly leading to an increase in quality of life.
  Interventions: Device: Transcutaneous Pulsed Electrical Stimulation (Device: WL-2103A)
- Trial Arm 2 (Experimental): Participants and experimenters are blinded. The aim of this study is to determine whether a battery-operated portable device (current adjustable) attached to the outer ears (tragus) makes one more likely to improve on their sleep and quality of daily life. Investigators believe this device encourages increases in vagal tone associated with increases in baroreflex sensitivity, improving sleep and possibly leading to an increase in quality of life.
  Interventions: Device: Transcutaneous Pulsed Electrical Stimulation (Device: WL-2103A)

INTERVENTIONS:
Device: Transcutaneous Pulsed Electrical Stimulation (Device: WL-2103A) — The Transcutaneous Electrical Nerve Stimulator (TENS) creates electrical impulses from a 9VDC-battery whose continuous intensity rate can be controlled by the user. The alligator clip with 2 electrodes is placed on the tragus part of the ear (shown to be 45% innervated via auricular vagus nerve) to stimulate the vagus nerve with an adjustable peak intensity (0-80mA), a frequency of 2 - 250Hz and a pulse width of 30-260 µsec. The vagus nerve contains a mixture of different types of nerve fibres, which are organized into bundles (fascicles). The fibres vary in diameter and conduction velocity, with A-type fibres the largest and fastest and C-type fibres the smallest and slowest, with B-type fibres intermediate. During nerve stimulation, fibres are activated in order of size from the largest (A-type) to the smallest (C-type). It has been suggested that A-type fibres are mainly activated during the stimulation via auricular vagus nerve.
  Other Names: Transcutaneous auricular vagal nerve stimulator; Transcutaneous Electrical Nerve Stimulator

SUMMARY:
Participants will be chosen at random to receive a 30-minute stimulation of a specialized nerve (called a vagus nerve). The aim of this study is to determine whether a battery-operated portable device (current adjustable) attached to the outer ears (tragus) makes one more likely to improve on their sleep and quality of daily life. Participants will visit the lab on 2 occasions (one with a stimulating device and one without), 3 weeks apart for detailed instruction on setting up the ear stimulation and sleep kit in their home. Researchers will compare the sleep results from a PSG sleep device from the 2 sessions to determine the effect, if any on sleep.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a 30-minute stimulation of the vagus nerve at the site of the tragus area of the outer ear, helps to improve sleep efficiency in healthy participants. The vagus nerve protects the heart and vital organs, by feeding back information to the brain, and subsequently mounting a protective response. The aim is to identify any potential benefits of a device to boost function of the vagus nerve.

The battery-operated portable electro-stimulator (sham, or active) (Transcutaneous auricular vagal nerve stimulation) is designed to be attached to the outer ear. The Transcutaneous Electrical Nerve Stimulator (TENS) (Model WL-2103A): creates electrical impulses from a 9VDC-battery whose continuous intensity rate can be controlled by the user. The alligator clip with 2 electrodes is placed on the tragus part of the ear (shown to be 45% innervated via auricular vagus nerve) to stimulate the vagus nerve with an adjustable peak intensity (0-80mA), a frequency of 2 - 250Hz and a pulse width of 30-260 micro-sec. The vagus nerve contains a mixture of different types of nerve fibres, which are organized into bundles (fascicles). The fibres vary in diameter and conduction velocity, with A-type fibres the largest and fastest and C-type fibres the smallest and slowest, with B-type fibres intermediate. During nerve stimulation, fibres are activated in order of size from the largest (A-type) to the smallest (C-type). It has been suggested that A-type fibres are mainly activated during the stimulation via auricular vagus nerve. It has been shown that a decrease in sympathetic activity and increase of parasympathetic modulation of the heart (controlled by the vagus nerve) creates the transition from wake to sleep states. Thus, stimulating the vagus nerve may maintain a balance of the autonomic nervous system and therefore, affect the quality of sleep.

The self-instrumented sleep evaluation device is a polysomnography (PSG) level 2 + ECG Prodigy Sleep System consisting of a chest mounted unit (CMU) that records heart-rate (ECG), breathing-rate (nasal cannula), chest and stomach movements, and leg movements. The head mounted unit (HMU) measures electroencephalogram (EEG) of the frontal lobe, eye and chin movements. The wrist unit records blood oxygen saturation (SpO2) and pulse rate. All the wearable devices sends the specific data to the table-top tablet (TTU) via Bluetooth. The system uses secured web-based PSG to analyze the EEG, electrooculogram (EOC), ECG, electromyogram, accelerometry, acoustic signals, nasal airflow, thoracic and abdomen respiratory effect, pulse rate and oxy-hemoglobin saturation. All results are scored using Michele Sleep Scoring System to create necessary files showing all the stages of sleep (N1, N2, N3, REM) including sleep length, desaturation and efficiency.

40-50 Participants will be asked to attend five study visits over a 1-2 month period:

1. Laboratory visit 1: Informed consent, screening (~ 1 hour)
2. Laboratory visit 2: Assessment of neuromodulation stimulation level using the lab stimulation device and demonstration of how-to self-instrument the Cerebra Sleep monitoring kit at their personal residence for 4 nights consecutively. Participants will be assigned to either a sham, or active stim device to self-administer and given the sleep questionnaires for each night. (~ 2 hours)
3. Laboratory visit 3: Return the equipment and questionnaires and de-brief on the past 4 nights (~ 30 mins)
4. Laboratory visit 4: (after 21-day washout period): Re-assessment of neuromodulation stimulation level and re-issue of a sleep kit. (~ 2 hours)
5. Laboratory visit 5: Return the equipment and debrief on the past 4 nights. (~30 mins)

During the laboratory visits, participants will be trained on how to complete a full self-instrumentation using the sleep unit. For the ear neuro-stimulator, participants will respond to the tester's prompts as they experience increases in the level of stimulation. Participants will then be chosen at random to receive either the 30 minutes of outer ear stimulation, or no stimulation since the final setting of the neuro-stimulator will not be observable.

The analysis will be conducted using a two-tailed, two sample t-test on the first intervention to determine there were no significant differences within the 2 groups (sham, or active). T-test for differences between the two groups.

All the sleep data will be encrypted and transferred to a secure database and all hard copied data will be separated from identifiers into a locked file storage system.

Once the study is finished, the participants will have the option to view individual results.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 and < 50 years.
* In good health with no evidence of medical problems.
* Ability to provide informed consent and willingness to comply with the study procedures.
* Ability to use a battery operated electro-stimulating device attached to your ears for 30 minutes.
* Ability to breathe through the nose comfortably and wear a sleep monitoring device.

Exclusion Criteria:

* Obesity (BMI > 40 kg/m2).
* Known history of heart, lung, kidney, or liver disease.
* Diagnosis of asthma or sleep apnea.
* Diagnosis of diabetes.
* Current smoker.
* Pregnancy or lactation due to the location of the sleep devices.
* Resting heart rate > 120 bpm.
* Systolic BP > 150, diastolic BP > 90.
* Presence of any other condition that, in the opinion of the PI, makes the individual unsuitable for participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Quality Evaluated by Polysomnography | 4 weeks
  Investigators believe this device encourages increases in vagal tone associated with increases in baroreflex sensitivity, improving sleep and possibly leading to an increase in quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Unviersity of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided